CLINICAL TRIAL: NCT01629563
Title: A Phase III, Multicentre, Randomized, Double-blind Clinical Study, Investigating the Efficacy and Safety of Repeated 12-week Courses of Daily 5mg or 10mg Doses of PGL4001 for the Long-term Management of Symptomatic Uterine Fibroids
Brief Title: PGL4001 Efficacy Assessment in Reduction of Symptoms Due to Uterine Leiomyomata
Acronym: PEARLIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PregLem SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGL11-006
Record Dates: First submitted 2012-06-19; First posted 2012-06-27 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ulipristal acetate (PGL4001) 5mg (Experimental): All subjects will be asked to take a 150mg size tablet (PGL4001 5mg or matching placebo: placebo 5) orally daily for repeated periods 84 days. The first treatment course will start on the first 4 days of menstruation and will be orally administered, once daily (1 tablet of 150mg size), for 84 days. The following three treatment courses should be started in the first two days of a menstrual period.
  Interventions: Drug: PGL4001 5 mg
- Ulipristal acetate (PGL4001) 10mg (Experimental): All subjects will be asked to take a 300mg size tablet (PGL4001 10mg or matching placebo: placebo 10 ) orally daily for repeated periods 84 days. The first treatment course will start on the first 4 days of menstruation and will be orally administered, once daily (1 tablet of 300mg size), for 84 days. The following three treatment courses should be started in the first two days of a menstrual period.
  Interventions: Drug: PGL4001 10 mg

INTERVENTIONS:
Drug: PGL4001 5 mg — PGL4001 5 mg daily administration
  Other Names: Ulipristal Acetate, Esmya
  Arms: Ulipristal acetate (PGL4001) 5mg
Drug: PGL4001 10 mg — PGL4001 10mg daily administration
  Other Names: Ulipristal Acetate
  Arms: Ulipristal acetate (PGL4001) 10mg

SUMMARY:
Phase III, multicentre, randomized, double-blind, parallel group, long-term study investigating the efficacy and safety of the 5mg and 10mg doses of PGL4001 for the treatment of uterine myoma.

DETAILED DESCRIPTION:
The target population is composed of pre-menopausal women with symptomatic uterine myoma(s) characterised by heavy bleeding.The main objective of this study is to assess the sustained efficacy and safety of long term on-off treatment with PGL4001 5 or 10mg doses on uterine bleeding, myoma size, pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Be a pre-menopausal woman between 18 and 50 years inclusive.
* Have a Body Mass Index (BMI) ≥ 18 and ≤ 40.
* Have FSH levels ≤ 20 mIU/mL
* Have excessive uterine bleeding due to myoma.
* Have regular menstrual cycles
* Have a myomatous uterus < 16 weeks with at least one myoma ≥ 3 cm in diameter.
* If of childbearing potential the subject must be practicing a non-hormonal method of contraception.

Exclusion Criteria:

* Has a history of or current uterine, cervical, ovarian or breast cancer.
* Has a history of or current endometrium atypical hyperplasia or adenocarcinoma.
* Has a known severe coagulation disorder.
* Has a history of or current treatment for myoma with a Selective Progesterone Receptor Modulator (SPRM).
* Has abnormal hepatic function at study entry.
* Has a positive pregnancy test, is nursing or planning a pregnancy during the course of the study.
* Has a current (within twelve months) problem with alcohol or drug abuse.
* Is currently enrolled in an investigational drug or device study or has participated in such a study within the last 30 days.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 451 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Arrigada, MD, Study Director — PregLem SA
Locations (48):
- Belgium (4):
  - Cliniques Universitaires Saint-Luc Gynécologie-Obstétrique, Brussels
  - UZ Leuven Campus Gasthuisberg, Leuven
  - CHU de Liège, CHR de la Citadelle Gynécologie-Obstétrique, Liège
  - CHU Mont-Godinne, Yvoir
- Czechia (7):
  - Centrum ambulantni gynekologie a primarni pece, Brno
  - FN Brno Gynekologicko - porodnická klinika, Brno
  - Sanatorium SANUS, Hradec Králové
  - Nemocnice Jihlava Gynekologicko - porodnicke oddeleni, Jihlava
  - G-CENTRUM Olomouc s.r.o., Olomouc
  - FN Olomouc, Porodnicko-Gynekologicka klinika, Olomouc
  - Femina Sana, s.r.o., Prague
- France (3):
  - Hôpital Bicêtre - APHP, Le Kremlin-Bicêtre
  - Hôpital Bichat, Service de Gynécologie Obstétrique, Paris
  - CHU Bretonneau Service de Gynécologie Obstétrique, Tours
- Germany (5):
  - Private practice, Hamburg
  - Medizinische Hochschule Hannover Klinik für Frauenheilkunde und Geburtshilfe, Hanover
  - Frauenarztpraxis, Hessen
  - Praxis für Frauenheilkunde, Klinische Forschung und Weiterbildung, Magdeburg
  - Technische Universität München, München
- Hungary (7):
  - Rethy Pal Korhaz és Rendelointezet Szuleszeti es Nogyogyaszati Osztaly, Békéscsaba
  - Institution Robert Karoly Maganklinika, Budapest
  - Szent Anna Szuleszeti, Nogyogyaszati es Ultrahang Maganrendelo, Debrecen
  - Josa Andras Oktatokorhaz, Nyíregyháza
  - Szuleszeti es Nogyogyaszati Osztaly, Szentes
  - Fejer Megyei Szent Gyorgy Korhaz Szuleszeti es Nogyogyaszati Osztaly, Székesfehérvár
  - Sandor Dent Bt., Szolnok
- Italy (2):
  - Dipartimento di Ostetricia e Ginecologia, Università degli Studi di Catanzaro "Magna Graecia", Catanzaro
  - Policlinico Universitario "Agostino Gemelli", Roma
- Latvia (3):
  - Riga 1. hospital, Riga
  - Latvian Medical Marine Center, Riga
  - Medical Company "ARS", Riga
- Lithuania (4):
  - Saules Family Medicine Center, Kaunas
  - Family Medicine Centre"Seimos Gydytojas", Vilnius
  - Private Clinic "Maxmeda", Vilnius
  - Private Clinic "Kardiolita", Vilnius
- Romania (6):
  - Centrul Medical SANA SRL, Bucharest
  - Quantum Medical Center SRL Obstetrica-Ginecologie, Bucharest
  - Fortis Medical Center SRL Obstetrica Ginecologie, Bucharest
  - Spitalul Clinic Dr. I.Cantacuzino sectia Obstetrica-Ginecologie, Bucharest
  - Centrul Medical EUROMED SRL, Departamentul de Obtetrica/Ginecologie, Bucharest
  - Spitalul Clinic de Obstetrica, Iași
- Ukraine (3):
  - Kharkiv City Perinatal Center Gynaecological Department #1, Kharkiv
  - Municipal Institution "Maternity Hospital #1" City Center of family planning, Odesa
  - Maternity Hospital#4 Department of Gynaecology, Zaporizhzhya
- United Kingdom (4):
  - MRC Centre for Reproductive Health University of Edinburgh, Edinburgh
  - North Middlesex University Hospital NHS Trust, London
  - Women's Health, Royal Victoria Infirmary, Newcastle upon Tyne
  - Norfolk & Norwich University Hospital, Norwich

REFERENCES:
- [Derived] Donnez J, Donnez O, Matule D, Ahrendt HJ, Hudecek R, Zatik J, Kasilovskiene Z, Dumitrascu MC, Fernandez H, Barlow DH, Bouchard P, Fauser BC, Bestel E, Loumaye E. Long-term medical management of uterine fibroids with ulipristal acetate. Fertil Steril. 2016 Jan;105(1):165-173.e4. doi: 10.1016/j.fertnstert.2015.09.032. Epub 2015 Oct 23. PMID 26477496
- [Derived] Donnez J, Hudecek R, Donnez O, Matule D, Arhendt HJ, Zatik J, Kasilovskiene Z, Dumitrascu MC, Fernandez H, Barlow DH, Bouchard P, Fauser BC, Bestel E, Terrill P, Osterloh I, Loumaye E. Efficacy and safety of repeated use of ulipristal acetate in uterine fibroids. Fertil Steril. 2015 Feb;103(2):519-27.e3. doi: 10.1016/j.fertnstert.2014.10.038. Epub 2014 Dec 24. PMID 25542821

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ulipristal Acetate (PGL4001) 5mg | Ulipristal Acetate (PGL4001) 10mg
Started (FAS population analysed As Randomised, Safety population analysed As Treated) | 228 | 223 (2 subjects randomised to 10mg received 5mg treatment in error (FAS 1: 10mg, Safety Set: 5mg))
Safety Population | 230 | 221
Started Treatment Course 2 | 213 | 207
Started Treatment Course 3 | 191 | 190
Started Treatment Course 4 | 178 | 176
Completed | 167 | 170
Not Completed | 61 | 53
Not completed — Adverse Event | 16 | 16
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 27 | 20
Not completed — surgery | 0 | 3
Not completed — Lack of return of menses | 12 | 7
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set 1(all subjects who received study treatment at least once for treatment course 1) (treament group as randomised)
Groups:
- Total: Total of all reporting groups
Arm/Group | Ulipristal Acetate (PGL4001) 5mg | Ulipristal Acetate (PGL4001) 10mg | Total
Number analyzed (Participants) | 228 | 223 | 451
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 228 | 223 | 451
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (5.4) | 41.4 (5.1) | 41.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 223 | 451
  Male | 0 | 0 | 0
Total volume of the 3 largest myoma [Median (Inter-Quartile Range); unit: cm3] — total volume of the three largest myomas (length, height and depth measured using transvaginal ultrasound, volume estimated by applying the equation for the volume of an ellipsoid (length × height × depth × π/6))
  cm3 | 42.6 [24.0 to 94.2] | 43.6 [27.3 to 117.3] | 43.3 [25.1 to 102.1]
Pain Assessment (Visual Analogue Scale) [Median (Inter-Quartile Range); unit: units on a scale] — Pain was assessed using a visual analogue scale (VAS) ranging from 0 to 100 with higher score indicating more severe pain.
  units on a scale | 39.0 [15.6 to 62] | 43.0 [19.0 to 67.0] | 40.5 [17.0 to 64.0]
Uterine Fibroid Symptom Quality of Life Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — Quality of Life was assessed using a validated questionnaire measuring uterine fibroid sympotom severity (UFSQoL) where lower scores indicate fewer symptoms and where a level of 23 has been reported for healthy subjects (scale 0-100).
  Total score for health related QoL (HRQL) ranges from 0 to 100 with higher score indicating better quality of Life.
  units on a scale
    Symptom Severity (UFSQoL) | 50.0 [37.5 to 62.5] | 50.0 [37.5 to 62.5] | 50.0 [37.5 to 62.5]
    Health related Quality of Life (HRQL) | 56.9 [42.2 to 75.9] | 55.2 [41.4 to 71.6] | 56.0 [41.4 to 73.3]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Are in Amenorrhea at the End of All Four Treatment Courses
Description: Amenorrhoea was defined as no more than 1 day of spotting within a 35 day interval. Subjects need to be in amenorrhoea at the end of all four treatment courses, i.e for at least 4x35 days.
Time Frame: 18 months study duration per subject (4 3-month intermittent treatment courses)
Population: Full Analysis Set 1 (subjects who received study treatment at least once for treatment course 1) (subjects with missing values were excluded from analysis)
Measure: Number; unit: percentage of subjects
Arm/Group | Ulipristal Acetate (PGL4001) 5mg | Ulipristal Acetate (PGL4001) 10mg
Number analyzed (Participants) | 195 | 185
percentage of subjects | 48.7 | 60.5

2. Secondary Outcome: Percentage of Subjects Who Were in Amenorrhea at the End of Treatment Course 4
Description: Amenorrhoea was defined as no more than 1 day of spotting within a 35 day interval.
Time Frame: After 18 months
Population: Full Analysis Set 1 (all subjects who received study treatment once for treatment course 1) (subjects with missing values were excluded from analysis)
Measure: Number; unit: percentage of participants
Arm/Group | Ulipristal Acetate (PGL4001) 5mg | Ulipristal Acetate (PGL4001) 10mg
Number analyzed (Participants) | 227 | 220
percentage of participants | 69.6 | 74.5

3. Secondary Outcome: Percentage of Subjects With Controlled Bleeding at the End of All 4 Treatment Courses
Description: Controlled bleeding was defined as no episodes of heavy bleeding and a maximum of 8 days of bleeding during the last 56 days of a treatment course.
  Subjects need to be in controlled bleeding at the end of all 4 treatment courses i.e. for at least 4x56 days.
Time Frame: After 18 months
Population: Full analysis set 1 (all subject who received study treatment at least once for treatment course 1) (subjects with missing values were excluded from analysis)
Measure: Number; unit: percentage of participants
Arm/Group | Ulipristal Acetate (PGL4001) 5mg | Ulipristal Acetate (PGL4001) 10mg
Number analyzed (Participants) | 158 | 146
percentage of participants | 67.1 | 71.9

4. Secondary Outcome: Percentage of Change From Baseline to End of Treatment Course 4 in the Total Volume of the 3 Largest Fibroids
Description: For the 3 largest myomas at baseline and the 3 largest myomas at the end of treatment course 4 identified by transvaginal ultrasound, length, height and depth were measured and the volume was estimated by applying the equation for the voulme of an ellipsoid (length x height x depht x π/6).
  Subjects were exposed to 4 3-month intermittent courses.
Time Frame: After 18 months
Population: Full Analysis Set 1 (all subjects who received study treatment at least once for treatment course 1) (subjects with missing values were excluded from analysis)
Measure: Median (Inter-Quartile Range); unit: percentage of change from baseline
Arm/Group | Ulipristal Acetate (PGL4001) 5mg | Ulipristal Acetate (PGL4001) 10mg
Number analyzed (Participants) | 160 | 159
percentage of change from baseline | -67.0 [-85.6 to -35.1] | -70.4 [-88.0 to -41.7]

5. Secondary Outcome: Percentage of Change From Baseline to End of Treatment Course 4 in Quality of Life (Uterine Fibroid Symptom Severity (UFSQoL)
Description: Quality of Life was assessed using a validated questionnaire measuring uterine fibroid symptom severity (UFSQoL) where lower scores indicate fewer symtoms and where a level of 23 has been reported for healthy subject (scale 0-100).
  Subjects were exposed to 4 3-month intermittent courses.
Time Frame: After 18 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage of change from baseline
Arm/Group | Ulipristal Acetate (PGL4001) 5mg | Ulipristal Acetate (PGL4001) 10mg
Number analyzed (Participants) | 137 | 137
percentage of change from baseline | -31.25 [-46.88 to -12.50] | -28.13 [-43.75 to -18.75]

6. Secondary Outcome: Percentage of Change From Baseline to End of Treatment Course 4 in Quality of Life -Uterine Fibroid Health Related Quality of Life (HRQL)
Description: Quality of Life was measured using a validated uterine fibroid symptom questionnaire. Total score for health related quality of Life (HRQL) range from 0 to 100 with higher scores indicating better Quality of Life.
  Subjects were exposed to 4 3-month intermittent courses.
Time Frame: 18 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage of change from baseline
Arm/Group | Ulipristal Acetate (PGL4001) 5mg | Ulipristal Acetate (PGL4001) 10mg
Number analyzed (Participants) | 136 | 138
percentage of change from baseline | 20.69 [6.47 to 35.34] | 15.52 [5.17 to 37.07]

7. Secondary Outcome: Percentage of Change From Baseline to End of Treatment Course 4 in Pain Using a Visual Analogue Scale (VAS)
Description: Pain was assessed using a Visual Analogue Scale (VAS) ranging from 0 to 100 with higher score indicating more severe pain.
  Subjects were exposed to 4 3-month intermittent courses.
Time Frame: After 18 months
Population: FAS1 (all subjects who received study treatment at least once for treatment course 1) (subjects with missing values were excluded from analysis)
Measure: Median (Inter-Quartile Range); unit: percentage of change from baseline
Arm/Group | Ulipristal Acetate (PGL4001) 5mg | Ulipristal Acetate (PGL4001) 10mg
Number analyzed (Participants) | 136 | 138
percentage of change from baseline | -20.0 [-46.1 to -0.5] | -23.0 [-52.0 to -1.0]

ADVERSE EVENTS:
Time Frame: Serious Adverse events were reported where the start date was on or after the first dose of study medication, up to the end of study follow-up (21 months on average).Other Adverse Events are summarised as on-treatment TEAEs.
Description: 2 subjects randomised to Ulipristal acetate 10 mg received 5 mg by mistake. They are included in the safety set according to treatment received.
  On-treatment TEAEs are events where the start date was on or after the first dose of study medication, up to and including 7 days after the last dose of study medication within each treatment course.
Arm/Group | Ulipristal Acetate (PGL4001) 5mg | Ulipristal Acetate (PGL4001) 10mg
Serious Adverse Events (participants affected / at risk) | 16/230 | 12/221
Other Adverse Events (participants affected / at risk) | 129/230 | 131/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ulipristal Acetate (PGL4001) 5mg (N=230) | Ulipristal Acetate (PGL4001) 10mg (N=221)
Menorrhagia (Reproductive system and breast disorders) | 4 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
arteriospam coronary (Cardiac disorders) | 0 | 1
tinnitus (Ear and labyrinth disorders) | 0 | 1
toxic nodular goitre (Endocrine disorders) | 1 | 0
abdominal pain (Gastrointestinal disorders) | 1 | 0
small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
accidental death (General disorders) | 1 | 0
homicide (General disorders) | 1 | 0
cholelithiasis (Hepatobiliary disorders) | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
breast hyperplasia (Reproductive system and breast disorders) | 0 | 1
endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
carpal tunnel syndrome (Nervous system disorders) | 0 | 1
bipolar disorder (Psychiatric disorders) | 1 | 0
urethral stenesis (Renal and urinary disorders) | 0 | 1
deep vein thrombosis (Vascular disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ulipristal Acetate (PGL4001) 5mg (N=230) | Ulipristal Acetate (PGL4001) 10mg (N=221)
headache (Nervous system disorders) | 31 | 30
hot flush (Reproductive system and breast disorders) | 18 | 23
influenza (Infections and infestations) | 12 | 10
nasopharyngitis (Infections and infestations) | 7 | 12
breast pain/breast tenderness/breast disconfort (Reproductive system and breast disorders) | 10 | 8
pelvic pain (Reproductive system and breast disorders) | 10 | 5
fatigue (General disorders) | 7 | 8
nausea (Gastrointestinal disorders) | 8 | 6
vaginal discharge (Reproductive system and breast disorders) | 5 | 7
back pain (Musculoskeletal and connective tissue disorders) | 5 | 6
abdominal pain (Gastrointestinal disorders) | 5 | 5
acne (Skin and subcutaneous tissue disorders) | 5 | 4
anxiety (Psychiatric disorders) | 5 | 4
aneamia (Blood and lymphatic system disorders) | 5 | 3
tonsillitis (Infections and infestations) | 4 | 5
hypertension (Vascular disorders) | 5 | 4
vertigo (Ear and labyrinth disorders) | 6 | 2
weight increased (Investigations) | 5 | 3
cystitis (Infections and infestations) | 3 | 5
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6
blood creatine phosphokinase increased (Investigations) | 5 | 2
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit to sponsor results communication for review 60 days prior to publication submission. If in the sponsor judgement, publication at a given time would hinder the sponsor's IP development, PI shall consider modifying the publication schedule. PI agrees to delete information identified by sponsor as confidential or defer publication to permit filing of patent application by the sponsor. Publication based on 1 site results shall not be made before the first muti-centre publication.